CLINICAL TRIAL: NCT05241795
Title: Crossover Effect of Knee and Ankle Joint Training on Knee Mechanics After Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial
Brief Title: Knee vs. Ankle Training on Knee Mechanics After ACLR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy Ali Hassan ElMeligie, Principal investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACL2122
Record Dates: First submitted 2022-02-05; First posted 2022-02-16 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: ACL Tear; ACL Sprain; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Knee exercises then Ankle exercises (Active Comparator): Patients will receive a rehabilitation protocol starting with knee training followed by ankle training.
  Interventions: Other: Knee then Ankle rehabilitation protocol
- Group B: Ankle exercises then Knee exercises (Experimental): Patients will receive a rehabilitation protocol starting with ankle training followed by knee training.
  Interventions: Other: Ankle then Knee rehabilitation protocol

INTERVENTIONS:
Other: Knee then Ankle rehabilitation protocol — Patients will start with knee exercise program that includes
  * Partial Squats: The exercise will be performed as 3 sets of 10 repetitions each day.
  * Toe Raises: The exercise will be performed as 3 sets of 10 repetitions each day.
  * Stationary bike will be used (10-15 minutes /day) when the patients can bend their knees at least 100 degrees, as cycling is considered as an excellent conditioning and building exercise for the quadriceps muscles. As the patient's ability to pedal the bike with the operative leg improved, the therapist will increase the resistance.
  * Hamstring exercises: After 6 weeks, the hamstring muscles will be exercised by the patient pulling the heel back producing a hamstring contraction.
  Then, Patients will start ankle exercises program that includes:
  * Standing calf raises
  * Foot lift
  * Ankle eversion exercises
  * Ankle Plantarflexion exercises
  Arms: Group A: Knee exercises then Ankle exercises
Other: Ankle then Knee rehabilitation protocol — Patients will start ankle exercises program that includes:
  * Standing calf raises
  * Foot lift
  * Ankle eversion exercises
  * Ankle Plantarflexion exercises
  Then, Patients will start with knee exercise program that includes
  * Partial Squats: The exercise will be performed as 3 sets of 10 repetitions each day.
  * Toe Raises: The exercise will be performed as 3 sets of 10 repetitions each day.
  * Stationary bike will be used (10-15 minutes /day) when the patients can bend their knees at least 100 degrees, as cycling is considered as an excellent conditioning and building exercise for the quadriceps muscles. As the patient's ability to pedal the bike with the operative leg improved, the therapist will increase the resistance.
  * Hamstring exercises: After 6 weeks, the hamstring muscles will be exercised by the patient pulling the heel back producing a hamstring contraction.
  Arms: Group B: Ankle exercises then Knee exercises

SUMMARY:
This study will be conducted to investigate if there is any difference between starting rehabilitation program after ACL reconstruction with knee joint training followed by ankle joint training and starting it with ankle joint training followed by knee joint training (crossover effect) on gait parameters of the knee joint.

ELIGIBILITY:
Inclusion Criteria:

* ACL reconstruction with a hamstring tendon autograft participated in this study.
* Score 7 on Tegner activity scale.

Exclusion Criteria:

* Patients with bilateral knee injury
* History of surgery or traumatic injury to the uninvolved lower extremity or to the hip or ankle of the involved lower extremity
* History of ACL reconstruction on the ipsilateral side and other knee ligament injuries requiring surgery.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-02-13 (Actual); Primary Completion 2022-07-21 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Knee joint flexion torques (Nm/kg) in the supporting (stance) phase at baseline and 6 weeks posttreatment | baseline and 6 weeks posttreatment
  Knee joint flexion torque (Nm/kg) in the supporting (stance) phase for each subject will be recorded using a 3D gait analysis system.
Change in Knee joint extension torques (Nm/kg) in the supporting (stance) phase at baseline and 6 weeks posttreatment | baseline and 6 weeks posttreatment
  Knee joint extension torque (Nm/kg) in the supporting (stance) phase for each subject will be recorded using a 3D gait analysis system.

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University Hospital, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication
Access Criteria: personal email: mohamed.magdy.pt@o6u.edu.eg